CLINICAL TRIAL: NCT03486080
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Safety and Efficacy Study of Dutogliptin in Combination With Filgrastim in Early Recovery Post-Myocardial Infarction
Brief Title: Study of Dutogliptin in Combination With Filgrastim in Post-Myocardial Infarction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Recardio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REC-DUT-002
Record Dates: First submitted 2018-03-12; First posted 2018-04-03 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Acute Myocardial Infarction; Acute Myocardial Ischemia; STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — dutogliptin; Filgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinded placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dutogliptin/filgrastim combination (Active Comparator): Twice daily SC injections of 60 mg dutogliptin tartrate for 14 days in combination with 10 µg/kg filgrastim injectable product for 5 days
  Interventions: Drug: Dutogliptin Tartrate; Drug: Filgrastim Injectable Product
- Placebo control (Placebo Comparator): Twice daily dutogliptin SC placebos for 14 days in combination with matching filgrastim SC placebos for 5 days
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Dutogliptin Tartrate — Active treatment
  Other Names: dutogliptin
  Arms: Dutogliptin/filgrastim combination
Drug: Filgrastim Injectable Product — Active treatment
  Other Names: filgrastim
  Arms: Dutogliptin/filgrastim combination
Drug: Placebos — placebo control
  Other Names: placebo
  Arms: Placebo control

SUMMARY:
A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Safety and Efficacy Study of Dutogliptin in Combination with Filgrastim in Early Recovery Post-Myocardial Infarction

DETAILED DESCRIPTION:
Dutogliptin 60 mg administered by twice daily subcutaneous (SC) injection for 14 days in combination with a fixed standard dose of filgrastim (10 µg/kg) administered SC daily for 5 days. This study will be conducted in adults with ST-elevation myocardial infarction (STEMI) with successful revascularization following percutaneous coronary intervention (PCI) and stent implantation.

Primary Objective

• To evaluate the safety and tolerability of dutogliptin in combination with filgrastim in subjects with STEMI compared with placebo

Secondary Objectives

* To assess preliminary efficacy of dutogliptin in combination with filgrastim in subjects with STEMI compared with placebo as determined by cardiac magnetic resonance imaging (cMRI)
* To determine the pharmacokinetics (PK) of dutogliptin in a subset of the study population
* To establish the pharmacodynamics (PD) of dutogliptin (plasma DPP4 activity) in a subset of the study population

Exploratory Objectives

* To examine the effects of dutogliptin in combination with filgrastim on:
* Change from baseline in plasma stromal cell-derived factor (SDF)-1a levels
* Change from baseline in plasma biomarkers, including N-terminal pro-b-type natriuretic peptide (NT-proBNP) and high sensitivity troponin

ELIGIBILITY:
Inclusion Criteria:

1. 1. Male or female born between 1933 and 2000.
2. Body weight <96 kg (212 lb).
3. Able to provide written informed consent, including signing and dating the informed consent form (ICF).
4. Diagnosis of STEMI (defined as new ST-segment elevation at the J point of at least 2 continuous leads of >2 mm [0.2 mV] in men or >1.5 mm [0.1 mV] in women in leads V2 and V3 OR >1 mm in any other contiguous precordial leads or the limb leads [for both men and women]) with PCI (bare metal or drug-eluting stent) and Thrombolysis in Myocardial Infarction flow grade 2 or 3 occurring >2 hours and <24 hours after symptom onset.
5. LVEF ≤45% obtained by cECHO performed within 36 hours post-stent placement.
6. Receiving standard medical therapy for post-MI treatment, according to local procedures and Principal Investigator discretion
7. Female subjects of childbearing potential must have a negative serum pregnancy test at Screening and an additional negative urine pregnancy test prior to the first dose of IMP unless regulated differently by national legislation.
8. Sexually active female subjects of childbearing potential (i.e., women who are not postmenopausal or who have not had a bilateral oophorectomy, hysterectomy, or tubal ligation) and all male subjects (who have not been surgically sterilized by vasectomy) must agree to use effective contraception during the study.

Exclusion criteria

1. Previous MI prior to Screening.
2. Complex peri/post-MI clinical course, including arrhythmias, cardiogenic shock, pulmonary edema requiring mechanical ventilation, or requirement for vasopressor medications.
3. Significant pre-existing cardiomyopathy with known LVEF ≤45% or moderate to severe mitral or aortic valvular disease.
4. Amyloidosis, hypertrophic obstructive cardiomyopathy, restrictive cardiomyopathy, or constrictive pericarditis.
5. Existing heart transplant.
6. Ventricular tachycardia or fibrillation not associated with an acute ischemic episode.
7. Uncontrolled hypertension (systolic >180 mmHg or diastolic >120 mmHg).
8. Treatment with any DPP4 inhibitors (e.g., alogliptin, linagliptin, vildagliptin, saxagliptin, sitagliptin) or G-CSF medication (e.g., filgrastim, lenograstim, pegfilgrastim, lipegfilgrastim) within 4 months prior to Randomization.
9. Contraindication to treatment with filgrastim, including known allergy to filgrastim or other G-CSF medication.
10. Anemia defined as hemoglobin <9 g/dL prior to Randomization.
11. Thrombocytosis (platelets >500 k/µL).
12. Known positive serology for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
13. Alanine aminotransferase (ALT) concentrations >3 times the upper limit of normal (ULN) or bilirubin >2 x ULN prior to Randomization, according to local laboratory assessments.
14. History of cirrhosis and Child-Pugh score B or C.
15. Current fever greater than 101.4 °F (38.6 °C) or recent systemic infection within 2 weeks prior to Randomization.
16. Contraindication to cMRI procedure, including prior implantable cardioverter defibrillator placement, known reaction to gadolinium, claustrophobia, non-MRI-compatible, cochlear implant, morbid obesity, or presence of ferromagnetic material including shunts, shrapnel, penile prostheses, or blood vessel coil.
17. Pregnant, planning to become pregnant, or nursing female subjects.
18. Autoimmune disease requiring immunosuppressive therapy or chronic steroid treatment >5 mg/day prednisolone or equivalent.
19. Significant renal impairment defined as estimated glomerular filtration rate <45 mL/min/1.73 m2, using the Chronic Kidney Disease Epidemiology Collaboration equation.
20. Active neoplasm requiring surgery, chemotherapy, or radiation within the prior 12 months (subjects with a history of malignancy who have undergone curative resection or otherwise not requiring treatment for at least 12 months prior to Screening with no detectable recurrence are allowed).
21. Malignant hematological disease, i.e., chronic myeloid leukemia or myelodysplastic syndrome.
22. History of cerebrovascular accident or transient ischemic attack in the past 6 months.
23. History of pneumonia in the last 4 weeks.
24. History of any significant medical or psychiatric disorder that in the opinion of the investigator would make the subject unsuitable for participation in the study.
25. Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) or treatment with an investigational biologic drug within 6 weeks prior to randomization.
26. Participation in another concurrent clinical trial involving a therapeutic intervention (participation in observational studies and/or registry studies is permitted).
27. Unable or unwilling to comply with the requirements of the study.
28. Subject and/or an immediate family member is an employee of the investigational site directly affiliated with this study, the sponsor or the contract research organization.
29. Considered by the investigator to be unsuitable to participate in the study for any other reason.
30. Persons who are in an institution as a result of an administrative or judicial order, or soldiers.
31. History of alcohol or drug abuse.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Safety assessment of the number of Grade 3 and 4 treatment emergent AEs or serious AEs (SAEs) as assessed by CTCAE v4.0.AEs (SAEs) as assessed by CTCAE v4.0. | 90 days
  Assess the tolerability of a combination of dutogliptin and filgrastim

SECONDARY OUTCOMES:
Cardiovascular efficacy LVEF | 90 days
  Left ventricular ejection fraction (%) by MRI
Cardiovascular efficacy LVESV | 90 days
  Left ventricular end systolic volume (mL) by MRI
Cardiovascular efficacy LVEDV | 90 days
  Left ventricular end diastolic volume (mL) by MRI
Cardiovascular tissue damage reduction | 90 days
  Infarct size (mm2)
Cardiovascular LFM | 90 days
  Left ventricular mass (mm2)
Cardiovascular motion | 90 days
  Regional wall motion (mm)
Pharmacokinetics (PK) | 14 days
  Assess the systemic exposure (dutogliptin AUC) of s.c. administered dutogliptin
Pharmacodynamics (PD) | 14 days
  Assess the PD effects (plasma DPP4 activity) of s.c. administered dutogliptin

CONTACTS AND LOCATIONS:
Overall Officials: Roman Schenk, MD, Study Chair — Recardio, Inc.
Locations (12):
- Austria (2):
  - Clinical department of Cardiology, Graz
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
- Algemeen Stedelijk Ziekenhuis Aalst, Aalst, Belgium
- Hungary (4):
  - Military Hospital, Budapest
  - Semmelweis Egyetem Városmajori Szív- és Érgyógyászati Klinika, Budapest
  - Debreceni Egyetem Kardiológiai és Szívsebészeti Klinika, Debrecen
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktatókórház, Miskolc
- Maasstad Ziekenhuis, Rotterdam, Netherlands
- Poland (4):
  - Nicolaus Copernicus University, Bydgoszcz
  - SPS Szpital Zachodni, Grodzisk Mazowiecki
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi ul. Pomorska 251, Lodz
  - Samodzielny Publiczny Szpital Wojewódzki im. Papieża Jana Pawła II, Zamość

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Recardio, Inc. Homepage — https://www.recardio.eu